CLINICAL TRIAL: NCT04174495
Title: Bone Fragility Evaluation by Dual X-Ray Absorptiometry (DXA) and CT-scan (vertebral Fracture and Scanographic Bone Attenuation Coefficient of the First Lumbar Vertebra SBAC-L1) in Obese Patients
Brief Title: Bone Fragility Evaluation in Obese Patients
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier de Toul Saint Charles (Unknown)
Responsible Party: Principal Investigator, Marine FAUNY, MD; Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2019PI216
Record Dates: First submitted 2019-11-16; First posted 2019-11-22 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity | interventions — Absorptiometry, Photon; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Obese patients followed at Nancy University Hospital
  Interventions: Diagnostic Test: DXA and CT-scan

INTERVENTIONS:
Diagnostic Test: DXA and CT-scan — DXA and CT-scan are usually performed during the following of these patients before bariatric surgery

SUMMARY:
This research will study the bone fragility in obese patients, on DXA and CT-scan, in a transversal study. The investigators want also to study the specific risk factors of bone fragility in these obese patients (relationship between body composition on whole body on DXA, fat mass and its location, lean mass, weight loss after surgery and SBAC-L1), to improve the bone screening.

ELIGIBILITY:
Inclusion Criteria:

* patients followed at Nancy university hospital for a bariatric surgery
* CT-scan and DXA performed before surgery, with maximum 1 year before the 2 exams

Exclusion Criteria:

* < 18 years
* Protected adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese patients followed before a bariatric surgery, at Nancy university hospital who performed a CT-scan and DXA, usually performed before surgery, with a delay which did not exceed 1 year before the 2 exams
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-02-23 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
scanographic bone attenuation coefficient of the first lumbar vertebra SBAC-L1 | November 2019-September 2020
  on axial section of the first lumbar vertebra, with a region of interest

SECONDARY OUTCOMES:
Vertebral fracture | November 2019-September 2020
  According Genant classification, on sagittal section of spine
DXA: T-score | November 2019-September 2020
  in standard deviation, on spine / hip / femoral neck / wrist
DXA: Bone mineral density BMD (spine, hip , femoral neck, wrist) | November 2019-September 2020
  in g/cm²
DXA: lean and fat mass | November 2019-September 2020
  in % and repartition of each

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy university hosiptal, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray TE, Williams D, Lee MJ. Osteoporosis, obesity, and sarcopenia on abdominal CT: a review of epidemiology, diagnostic criteria, and management strategies for the reporting radiologist. Abdom Radiol (NY). 2017 Sep;42(9):2376-2386. doi: 10.1007/s00261-017-1124-5. PMID 28386693
- [Background] Walsh JS, Vilaca T. Obesity, Type 2 Diabetes and Bone in Adults. Calcif Tissue Int. 2017 May;100(5):528-535. doi: 10.1007/s00223-016-0229-0. Epub 2017 Mar 9. PMID 28280846
- [Background] Hammoud E, Toumi H, Jacob C, Pinti A, Lespessailles E, El Hage R. Does the Severity of Obesity Influence Bone Mineral Density Values in Premenopausal Women? J Clin Densitom. 2021 Apr-Jun;24(2):225-232. doi: 10.1016/j.jocd.2019.04.006. Epub 2019 Apr 26. PMID 31109773
- [Background] Bauer JM, Cruz-Jentoft AJ, Fielding RA, Kanis JA, Reginster JY, Bruyere O, Cesari M, Chapurlat R, Al-Daghri N, Dennison E, Kaufman JM, Landi F, Laslop A, Locquet M, Maggi S, McCloskey E, Perna S, Rizzoli R, Rolland Y, Rondanelli M, Szulc P, Vellas B, Vlaskovska M, Cooper C. Is There Enough Evidence for Osteosarcopenic Obesity as a Distinct Entity? A Critical Literature Review. Calcif Tissue Int. 2019 Aug;105(2):109-124. doi: 10.1007/s00223-019-00561-w. Epub 2019 May 16. PMID 31098729
- [Background] Jammah AA. Endocrine and metabolic complications after bariatric surgery. Saudi J Gastroenterol. 2015 Sep-Oct;21(5):269-77. doi: 10.4103/1319-3767.164183. PMID 26458852
- [Background] Hong CS, Bergen MA, Watters TS. Transient osteoporosis of the hip after bariatric surgery. Arthroplast Today. 2018 Dec 7;5(1):32-37. doi: 10.1016/j.artd.2018.10.010. eCollection 2019 Mar. PMID 31020018
- [Background] Lespessailles E, Hammoud E, Toumi H, Ibrahim-Nasser N. Consequences of bariatric surgery on outcomes in rheumatic diseases. Arthritis Res Ther. 2019 Mar 28;21(1):83. doi: 10.1186/s13075-019-1869-z. PMID 30922375
- [Background] Santos D, Lopes T, Jesus P, Cruz S, Cordeiro A, Pereira S, Saboya C, Ramalho A. Bone Metabolism in Adolescents and Adults Undergoing Roux-En-Y Gastric Bypass: a Comparative Study. Obes Surg. 2019 Jul;29(7):2144-2150. doi: 10.1007/s11695-019-03797-5. PMID 30820885
- [Background] Geoffroy M, Charlot-Lambrecht I, Chrusciel J, Gaubil-Kaladjian I, Diaz-Cives A, Eschard JP, Salmon JH. Impact of Bariatric Surgery on Bone Mineral Density: Observational Study of 110 Patients Followed up in a Specialized Center for the Treatment of Obesity in France. Obes Surg. 2019 Jun;29(6):1765-1772. doi: 10.1007/s11695-019-03719-5. PMID 30734230
- [Background] Madsen LR, Espersen R, Ornstrup MJ, Jorgensen NR, Langdahl BL, Richelsen B. Bone Health in Patients with Type 2 Diabetes Treated by Roux-En-Y Gastric Bypass and the Role of Diabetes Remission. Obes Surg. 2019 Jun;29(6):1823-1831. doi: 10.1007/s11695-019-03753-3. PMID 30719648
- [Background] Axelsson KF, Werling M, Eliasson B, Szabo E, Naslund I, Wedel H, Lundh D, Lorentzon M. Fracture Risk After Gastric Bypass Surgery: A Retrospective Cohort Study. J Bone Miner Res. 2018 Dec;33(12):2122-2131. doi: 10.1002/jbmr.3553. Epub 2018 Aug 13. PMID 30011091
- [Background] Mesureur L, Arvanitakis M. Metabolic and nutritional complications of bariatric surgery : a review. Acta Gastroenterol Belg. 2017 Oct-Dec;80(4):515-525. PMID 29560648
- [Background] Kalani A, Bami H, Tiboni M, Jaeschke R, Adachi JD, Lau AN. The effect of bariatric surgery on serum 25-OH vitamin D levels: a systematic review and meta-analysis. Obes Sci Pract. 2017 Jun 27;3(3):319-332. doi: 10.1002/osp4.113. eCollection 2017 Sep. PMID 29071108
- [Background] Cook FJ, Khanna I, Giordano J, Matarese L, Hudson S. LONG-TERM BONE HEALTH AFTER ROUX-EN-Y GASTRIC BYPASS: A PILOT STUDY. Endocr Pract. 2017 Sep;23(9):1077-1084. doi: 10.4158/EP171823.OR. Epub 2017 Jul 6. PMID 28683234
- [Background] Shanbhogue VV, Stoving RK, Frederiksen KH, Hanson S, Brixen K, Gram J, Jorgensen NR, Hansen S. Bone structural changes after gastric bypass surgery evaluated by HR-pQCT: a two-year longitudinal study. Eur J Endocrinol. 2017 Jun;176(6):685-693. doi: 10.1530/EJE-17-0014. Epub 2017 Mar 13. PMID 28289103
- [Background] Yu EW, Lee MP, Landon JE, Lindeman KG, Kim SC. Fracture Risk After Bariatric Surgery: Roux-en-Y Gastric Bypass Versus Adjustable Gastric Banding. J Bone Miner Res. 2017 Jun;32(6):1229-1236. doi: 10.1002/jbmr.3101. Epub 2017 Mar 20. PMID 28251687
- [Background] Pickhardt PJ, Lee LJ, del Rio AM, Lauder T, Bruce RJ, Summers RM, Pooler BD, Binkley N. Simultaneous screening for osteoporosis at CT colonography: bone mineral density assessment using MDCT attenuation techniques compared with the DXA reference standard. J Bone Miner Res. 2011 Sep;26(9):2194-203. doi: 10.1002/jbmr.428. PMID 21590738
- [Background] Fauny M, Bauer E, Albuisson E, Perrier-Cornet J, Deibener J, Chabot F, Mandry D, Huttin O, Chary-Valckenaere I, Loeuille D. Vertebral fracture prevalence and measurement of the scanographic bone attenuation coefficient on CT-scan in patients with systemic sclerosis. Rheumatol Int. 2018 Oct;38(10):1901-1910. doi: 10.1007/s00296-018-4139-5. Epub 2018 Aug 21. PMID 30132216
- [Background] Perrier-Cornet J, Omorou AY, Fauny M, Loeuille D, Chary-Valckenaere I. Opportunistic screening for osteoporosis using thoraco-abdomino-pelvic CT-scan assessing the vertebral density in rheumatoid arthritis patients. Osteoporos Int. 2019 Jun;30(6):1215-1222. doi: 10.1007/s00198-019-04931-w. Epub 2019 Mar 13. PMID 30868182
- [Background] Fauny M, Albuisson E, Bauer E, Perrier-Cornet J, Chary-Valckenaere I, Loeuille D. Study of vertebral fracture and Scanographic Bone Attenuation Coefficient in rheumatoid arthritis and ankylosing spondylitis vs. controls. Sci Rep. 2019 Sep 16;9(1):13323. doi: 10.1038/s41598-019-49712-x. PMID 31527613